CLINICAL TRIAL: NCT06363500
Title: Characterization of HIV-1 Reservoirs in HIV+ Adolescents
Brief Title: Characterization of HIV-1 Reservoirs in HIV-1 Non-B Infected Adolescents on ART in Cameroon
Acronym: AVIR
Status: Completed | Type: Observational
Sponsor: Chantal Biya International Reference Centre for Research on Prevention and Management of HIV/AIDS (Other Government)
Responsible Party: Principal Investigator, Judith Ndongo Embola Torimiro, Researcher, Chantal Biya International Reference Centre for Research on Prevention and Management of HIV/AIDS
Other Study IDs: ChantalIRCB
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Characterization of HIV Reservoirs in Adolescents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA samples extracted from PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non applicable — Only blood sample collection

SUMMARY:
Background: Combination antiretroviral therapy (cART) can bring HIV-1 in blood plasma to level undetectable by standard tests and allow a near-normal life expectancy for HIV-infected individuals. Unfortunately, cART is not curative, as within a few weeks of treatment cessation, HIV viremia in most patients rebounds except for rare elite or post-treatment controllers of viremia. The primary source of this rebound is the highly stable reservoir of latent yet replication-competent HIV-1 proviruses integrated into the genomic DNA of resting memory CD4+ T cells. To achieve a cure for HIV, understanding the cell reservoir environment is of paramount importance. The size and nature of viral reservoir might vary per timing of therapy, therapeutic response, ART duration, and immune response. Mechanisms of reservoir maintenance generally depend on levels/type of immune recognition, dynamics of viral persistence are different between pediatric and adult populations, owing to, but not limited to, types/numbers of target cells, efficiency in clearing HIV-infected cells, plasma viremia and HIV drug resistance patterns. This difference could become more evident as these children grow toward adolescence (increasing population due to ART benefits), a stage during which suboptimal adherence is frequent, leading to viral rebound and archiving of resistant patterns.

Objectives: We plan to conduct a cross sectional study with the aim to characterize HIV reservoirs and their variability according to virological and immunological profiles of non-B HIV-1 vertically infected adolescents receiving antiretroviral therapy. Specifically, we shall (1) evaluate the size of HIV reservoir; (2) Determine HIV-1 genetic variability and drug resistance in cellular reservoirs; (3) Characterize immune activation/inflammation of HIV infected adolescents.

Methods: We plan to conduct an observational and comparative study involving 90 HIV-1 non-B infected adolescents aged 10-19 years vertically infected, have been on ART for at least 12 months selected from a cohort of the ongoing EDCTP-READY study; intravenous blood will be collected for CD4/CD8 count, plasmatic viral load, PBMCs isolation, immune activation/inflammatory markers, genotyping and Viral reservoir quantification. We will as well recruit a group of 30 HIV-negative adolescents as control for immunological profiling.

Overall impact: Our findings will help in advancing knowledge on HIV reservoir, in terms of size and genetic variability in adolescents living with HIV (ADLHIV). Such evidence will also help in understanding the effects of ART timing and duration on the size of reservoirs among ADLHIV, a unique population from whom findings generated will largely contribute in designing functional cure strategies in this vulnerable population.

DETAILED DESCRIPTION:
Title: Characterization of Viral Reservoirs among HIV-1 non-B Vertically Infected Adolescents receiving Antiretroviral Therapy in Cameroon.

Acronym: AVIR-study, Adolescent viral reservoir

Importance and relevance Sub-Saharan Africa (SSA) is disproportionally affected with HIV/AIDS, with close to 70% of the global epidemics. With the highest burden of paediatric HIV infections, about nine out of every 10 children living with HIV found in the SSA region(1, 2). Adolescents and young people represent a growing share of people living with HIV worldwide. In 2019, about 1.7 million [1.1 million-2.4 million] adolescents between the ages of 10 and 19 were living with HIV worldwide representing about 5% of all people living with HIV, about 1.5 million [1.0 - 2.1 million] or 88% of HIV infected adolescent live in SSA. In 2019 alone, 460,000 [260,000-680,000] young people between the ages of 10 to 24 were newly infected with HIV, of whom 170,000 [53,000-340,000] were adolescents between the ages of 10 and 19. To compound this, most recent data indicate that only 27% of adolescent girls and 16% of adolescent boys aged 15-19 in Eastern and Southern Africa - the region most affected by HIV - have been tested for HIV in the past 12 months and received the result of the last test. The testing rates in West and Central Africa and South Asia are even lower. If current trends continue, hundreds of thousands more will become HIV-positive in the coming years, and without knowing their status, adolescents will miss out on life-saving treatment. Additionally, a large population of children infected with HIV perinatally over the last decade are growing into adolescence (3). Of the estimated 690,000 people who died of AIDS-related illnesses in 2019, 110,000 (or approximately 16%) of them were children under 20 years of age. (UNICEF global and regional trends, July 2020).

With the advent and scalability of Antiretroviral therapy (ART), there is a global decrease in AIDS-related deaths. As of the end of 2019, 25.4 million people were accessing antiretroviral therapy, representing 67% of all people living with HIV. However, only 53% of children living with HIV were receiving ART. Interestingly, about 94% of all children receiving ART are from SSA (4). In this context of continuous new HIV paediatric infections and increasing coverage in paediatric ART, the number of children living with HIV will increase, suggesting a higher likelihood of reaching adolescent age and even adulthood if treatment regimens remain fully effective in controlling HIV infection (3, 4). ADLHIV therefore constitutes an HIV population with growing health concerns and with very limited findings for generalizable best practices specific to this target population, especially in SSA.

Like several West and Central African countries, Cameroon is still faced with a generalized HIV epidemiology (2.7% prevalence) (5), with higher prevalence among pregnant women (5.7%) and HIV-exposed infants/children (5.8% [958/16,638] positivity at first PCR and 15% at the end of the PMTCT cascade) (6). As of June 2018, the national coverage of ART was 51.5% (281,083), which includes 12,362 children below 15 years of age (6). Regarding response to ART in Cameroon, we reported an overall rate of 79.4% viral suppression, with significant disparities across age ranges: 81.1% in adults, 75.6% in children, and only 53.3% in adolescent aged 10-19 years (7). Similar to UNAIDS reports, adolescents living with HIV (ADLHIV) represent the most vulnerable and underserved population in response to the epidemics(1, 5). For a safer growth toward adulthood, there is need to prioritize this population for the quest of innovative treatment strategies that ensure their well-being and their contribution for the development of SSA.

In spite of the unquestioned benefits of ART, there are limitations with current treatment strategies. Of note, the lifelong nature of current ART goes with challenges related adherence for most patients, ART-attributed toxicities and persisting immune dysfunction have significant health impairments, and HIV drug resistance (HIVDR) is increasing, mostly in SSA countries where most ART-experienced patients are living (8). There is a threat of an emerging new HIV epidemic, driven by HIVDR to existing antiretroviral. These challenges are particularly true for paediatric populations due to limited ART options, poor drug formulations, and increasing events of non-adherence as they grow toward adolescence. These challenges call for approaches toward HIV (functional) cure or remission, especially for the most vulnerable populations (i.e. ADLHIV) (7, 9).

Concepts underpinning the project including ideas and models or assumptions HIV-1 remission or eradication strategies aim to achieve viral remission in the absence of antiretroviral therapy (ART). The development of an HIV-1 cure remains challenging due to the latent reservoirs. The HIV-1 Latent Reservoir (LR) can be defined as the fraction of cells harbouring transcriptionally silent proviral DNA that are capable of producing infectious virions following activation(10). Resting memory CD4T cells are the primary host of the LR but HIV-1 infection in these cells is inefficient due their low co-receptor expression and inherent restrictions to reverse transcription (11, 12). Nevertheless, there is evidence that HIV-1 can infect resting CD4T cells directly or via cell-to-cell transmission, though infection in these cells is associated with slower replication kinetics (13). Alternatively, latency is established when a subset of infected, activated CD4T cells revert to a resting memory phenotype, effectively silencing viral gene expression whilst sustaining the proviral DNA long-term(14). The provirus is maintained in a quiescent state in these cells via host factors such as epigenetic suppression, depletion of transcription factors such as NF-κB and transcriptional interference due to integration into expressed genes, reviewed in more detail (15). Viral rebound from the LR following ART cessation is rapid, leading to detectable viremia within weeks of therapy interruption (16). Additionally, initiating ART early in infection is not sufficient to stop the formation of the LR, suggesting the LR is established and disseminated early (Chun et al., 1998; Whitney et al., 2014; Colby et al., 2018), even in vertically infected children that started ART soon after birth (17). The latent reservoir is stable despite years of suppressive ART and is the source of rebound viremia following therapy interruption. Latently infected cells therefore represent the principle barrier to an HIV- 1 cure and should be specifically targeted by novel treatment and eradication strategies.

The progress toward the development of a functional or sterilizing cure for HIV-1 has been significantly hindered by the presence of the LR. Currently, two people have been cured of HIV-1 infection, the so-called Berlin and London patients, who since receiving allogenic stem cell transplantations from CCR5?32/?32 donors, have consistently tested negative for viral rebound for over 10 and 2 years, respectively, without ART (18). In these cases, the infected cell pool was significantly depleted during pre- transplant conditioning and replaced with donor cells that are resistant to infection with R5-tropic virus due a large deletion in the CCR5 co-receptor (19). Due to the relative paucity of CCR5 ?32/?32 donors and the unique circumstances predetermining these cases, this type of cure is not feasible for widespread use, it does however emphasize the basic principle of HIV-1 cure; silence or eradicate the HIV-1 LR (20). Over the past decade, understanding of where and how HIV persists in individuals on ART has transformed substantially with evidence that virus persists in multiple cell types and tissue sites, and in both quiescent and proliferating long-lived latently infected cells. Thus, in the frame of a suppressive treatment, accurate estimates of the viral reservoir would help in a better mastering of viral persistence, which in turn might overcome existing barriers for achieving a cure(21).

Total HIV DNA is a reference biomarker that includes both integrated and unintegrated HIV DNA and reflects the global level of the viral reservoir. Importantly, Buzon et al. reported a statistical correlation between the time from HIV infection to treatment initiation and the total HIV DNA level after 10 years of continuous treatment in a cohort of adults first treated with early infection (22). In children, the HIV DNA level was markedly lower when viral control was achieved before the age of 1 year (23). By comparison with other markers, total HIV DNA has the advantage of easy quantification by standardized, sensitive, real- time PCR, including digital droplet PCR (ddPCR) (24).

Generalized immune activation is a hallmark of HIV-1 infection. In this state, a variety of immune cells show an increase in expression of activation, proliferation, and apoptotic markers, cellular turnover with aberrant cell cycle regulation, production of pro-inflammatory cytokines, and increased lymphoid tissue fibrosis (25). Immune activation is strongly associated with HIV-1 disease progression; for instance, T cell activation, as measured by expression of CD38 and HLA-DR, is more predictive of CD4+T cell depletion and shorter survival than is the plasma viral load (26, 27). Furthermore, the level of immune activation early in HIV-1 infection as measured by CD8+T cell activation predicts CD4+T cell loss independently of plasma HIV-1 RNA levels (28). Suppression of viral replication with effective antiretroviral treatment (ART) reduces immune activation, but even effective ART regimens are unable to reduce the levels of immune activation in HIV-infected individuals to levels seen in healthy individuals (25). HIV-infected children, even if successfully treated with ART, face a lifetime of elevated immune activation. Thus, evaluating the potential impact of chronic immune activation and inflammation on the developing immune system and on disease outcome in paediatric HIV infection is of particular importance. Recent studies showed that immune activation (HLA-DR, CD38) and exhaustion markers (Tim-3, PD-1, Lag-3) are strongly associated with reservoir size in ART- treated adults, thus it might be anticipated that minimizing the viral reservoir with early ART might, equally, minimize the level of immune activation and the non-AIDS 'ageing' diseases associated with persistent immune activation.

There is limited evidence in characterizing HIV reservoirs in West and Central African region, a geographical setting having a highest variability in circulating HIV-1 and HIV-2 strains (29, 30). For example, Cameroon, a zoonotic epicentre of HIV-1, is host to an extensively diverse landscape of HIV driven by the CRF02_AG recombinant, including most group M (sub-) subtypes, a vast array of URFs and CRFs, and group N, O, P and HIV-2 viruses(31-33). Thus, generating baseline data on the genotypic and quantitative profile of the viral reservoir across several HIV clades in setting like Cameroon would inform the design of optimal strategies for HIV cure. Considering the aforementioned vulnerability of adolescents with vertical infection and the limited knowledge on viral reservoirs and immune activation/inflammatory reaction in this population, evidence generated from this target will be highly complementary to current global efforts. Such evidence, generated in a context of high burden of co-infections (34, 35), might depict differential mechanisms of HIV persistence far from those reported in other parts of the World.

Preliminary work:

Within the frame of the ongoing EDCTP READY-Study, we have set up a cohort of 292 vertically infected adolescents (10-19 years) receiving ART in Cameroon. In this cohort, we reported a rate of 40% undetectable viral load (<40 copies/mL) after a median of 8 years of ART, about 20% immunological failure (CD4<250 cells/mm3) rate and less than 10% clinical failure (i.e. WHO stages III/IV) (36). This population offers a unique opportunity for understanding the size and nature of the reservoir, the variability of immune response/cytokine profiling, and the effect of viral subtype, treatment history (ART regimen and duration), gender disparities and adherence level on the control of viral reservoir.

AIM:

The aim of this study is to characterize HIV reservoirs and their variability according to virological and immunological profiles of vertically infected adolescents receiving antiretroviral therapy in Cameroon, and therefore, improve understanding of viral reservoirs and provide accurate and reliable data for HIV cure research.

Specific Objectives:

In this study, we shall: 1- Determine HIV-1 genetic variability and drug resistance in cellular reservoirs; 2- Characterize immune activation/inflammation in adolescents vertically infected with HIV-1; 3- Evaluate the size of HIV reservoir; 4- Evaluate the effect of antiretroviral therapy and immune response on the viral reservoir profile.

Materials and Methods Study design We plan to conduct an observational and comparative study among adolescent living with HIV and receiving ART in Cameroon. Participants will be selected and enrolled from an existing cohort of close to 300 vertically infected adolescents recruited for the EDCTP-READY study.

The EDCTP-READY-Study main objective was to evaluate treatment response, drug resistance and HIV-1 variability among adolescents on first- and second-line antiretroviral therapy in Cameroon (7). In this study, we recruited 296 HIV+ adolescents and compared the HIV-1 genotypic profile in circulating-RNA. Out of 30% (89/296) APHI experiencing virological failure (VL>1000 copies/mL).

Sampling method:

Blood samples will be collected from participants of EDCTP-READY study according to the eligibility criteria.

Eligibility criteria:

Inclusion criteria: Will be enrolled in the study, HIV+ adolescents aged 10-19 years old, vertically infected, have been on ART for at least 12 months, who provide their written assent and whose legal guardian provide written proxy-consent.

Non-inclusion criteria: Will not be considered for enrolment, HIV+ adolescent with incomplete ART history, HBV/HCV and malaria coinfections.

Exclusion criteria: Will be considered excluded from the study, any participant who decides freely to withdraw after had given consent or unable to give blood sample.

Sample size: The minimum sample size (N) of the study is 90 participants, calculated based on the following formula: N=p (1-p) (Zα2/α2); N = 0.02(1-0.02) (1.962/0.052) = 30 per arm (arm-A: VL<40 copies/mL; arm-B: VL 40-999 copies/mL; arm-C: viral load ≥1000 copies/mL). P is the prevalence of adolescents living with HIV in Cameroon with P=2% [3]; α being the risk agrees with α = 5%; Zα being the small gap with Zα = 1.96.

NB: A group of 30 HIV-negative adolescents will serve as control for immunological profiling.

All participants will be assigned a new identification number and data will be centralized in a password-protected computer at the International Reference Centre Chantal Biya (CIRCB) for research on HIV/AIDS prevention and management.

Study procedures and variables Procedures and timelines The present study requires 18 months to be completed: 3 months (month 1-3) for administration and ethics approval, 12 months (month 4 to 15) for enrolment of participants, sampling and laboratory analyses, 3 months (month 16 to 18) for data processing and reporting, see Gantt chart for more details.

Based on inclusion criteria, HIV+ adolescents case report forms will be selected from EDCTP-READY study and their legal guardian will be contacted. Assent and proxy-informed consent will be obtained from adolescents and legal guardian, respectively. Socio-demographic, clinical data and ART history will be assessed again for the period during enrolment in EDCTP-READY study. Then 90 or more HIV+ adolescents [30 per arm (arm-A: VL<40 copies/mL; arm-B: VL 40-999 copies/mL; arm-C: viral load ≥1000 copies/mL)] will be enrolled. A group of 30 HIV-negative adolescents will be enrolled to serve as control for immunological profiling. Intravenous blood (5ml x 2) will be collected by a trained phlebotomist for lab analyses including PBMCs isolation, plasma and buffy coat isolation, CD4/CD8 counts, plasmatic viral load (PVL), immune activation / inflammatory markers assessment, HIV-RNA and HIV-DNA genotyping, quantification of viral reservoirs.

HIV negative participants will be recruited at the CIRCB, this institution is a reference Centre for management of HIV infected individuals since 2006, and as such is renown reference centre for HIV testing. Base on this advantage, CIRCB organizes free HIV/HBV/HCV screening tests for several institutions and communities per year, therefore, a similar free testing campaign will be organized in a nearby secondary school and the present study will be presented to those fulfilling inclusion criteria. Potential participants will be invited at CIRCB with their legal guardian for enrolment.

Samples will be collected only once at enrolment as well as all relevant socio-demographic and clinical data. Samples will be transported to CIRCB the same day for PBMCs isolation, DNA, plasma and buffy coat isolation, CD4/CD8 counts and activation / inflammatory markers assessment using flow cytometry. Plasma will be collected and stored at -80oC for plasmatic viral load (PVL), genotyping, immune activation / inflammatory markers assessment using ELISA tests (or flow cytometry). HIV-DNA will be subsequently extracted from PBMCs and stored at -80oC; HIV-DNA will be shipped every three months to the department of experimental medicine, University of Rome Tor Vergata, Rome, Italy, for HIV viral reservoir quantification (see letter of collaboration in annex section).

Laboratory procedures CD4/CD8 count: CD4/CD8 measurements will be determined using flow cytometry machine as previously described (37).

Plasma viral load: Plasma viral load will be determined using m 2000rt Abbott real time system as previously described (38).

HIV-RNA extraction: ARN will be extracted from plasma samples using Qiamp viral RNA Mini Kit (Qiagen) as described by the manufacturer.

Pro-viral DNA extraction from buffy coat: Pro-viral DNA will be extracted using DNeasy blood and tissue extraction kit (Qiagen) as described by the manufacturer.

PBMCs isolation: PBMCs will be isolated by density gradient centrifugation using Ficoll using an in-house protocol.

HIV-DNA extraction from PBMCs: HIV-DNA will be extracted using QIAmp DNA Mini Kit (Qiagen) as described by the manufacturer.

HIV-1 Genes amplification and sequencing: Sanger Sequencing for HIV-1 drug resistance testing will be performed for adolescent experiencing virological failure an in-house protocol, as previously described by our research group(39). Reverse transcriptase DNA sequences will be analysed for drug resistance mutations using the Stanford University database genotypic resistance interpretation algorithm (www.stanford.edu).

Phylogenetic analysis: Neighbour Joining phylogenetic trees will be created using MEGA software (Kimura 2-parameter model, 200 bootstrap replications) and FigTree (40, 41).

Immune profiling: Both immune activation/inflammatory cytokines (IL-1, IL2,IL4, IL6, IL10, IL12 and TNF-alpha) will be assessed using commercial ELISA kits and flow cytometry.

Quantification of HIV viral reservoirs: viral reservoirs will be quantified using droplet digital PCR (ddPCR) as previously described. Of note, this quantification will be performed in the department of experimental medicine, University of Rome Tor Vergata, Rome, Italy as stated in the letter of collaboration found in annex of this proposal. A material transfer and a data sharing agreement will be signed between CIRCB and UTV prior to sample shipment to UTV. It is an in-house protocole for HIV-1 B subtype and will be adjusted for HIV-1 non-B subtypes expected from Cameroonian samples.

Data analysis Data collected during the study will be analyzed using SPSS software. Associated factors will be evaluated using multivariate logistic regression, with an estimate approach for the unbiased effect of different parameters. The data will be reported as median. Non-parametric tests will be used for data not normally distributed, comparisons of medians among different groups (virological success vs virological failure) will be performed by the U-Mann- Whitney test. Correlations will be made with Spearman test and p values less than 0.05 will be considered to be statistically significant.

Ethical considerations This study will be conducted according to the declaration of Helsinki on ethical principles for medical research involving human subjects. Ethical clearance will be obtained from the Cameroon National Ethics committee for research on human health. after an informed notice on the study, a written proxy-informed will be obtained from legal guardian, and a written assent will also be obtained from the participating HIV+ adolescent, without any coercion. Privacy and confidentiality will be ensured, through the use of unique identifiers and a password protected database and will be accessed only by authorized staff. Participants will be free to deliberately leave the study at any time, without any effect on their routine monitoring at the study clinic. Phlebotomy will be non-invasive (venipuncture) and will be performed by a trained nurse.

Quality assurance:

Our study team will include a quality assurance officer who will be responsible of all SOPs for the study protocol and will manage proficiency testing and data validation during the entire study.

Management of potential risks: The risks to the patients are minimal since the only procedure the volunteer is subjected to is venipuncture by a phlebotomist or physician. The venipuncture may be slightly painful, but is practically without risk of complication. The potential risks to subjects, none of which are likely to occur, may include momentary pain, bruising at the site or possible (but extremely unlikely) infection. If such complications arise, participant will be provided with emergency medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Consenting HIV+ Adolescents on ART

Exclusion Criteria:

* Insufficient blood for lab tests

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: HIV+ adolescents on antiretroviral treatment
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Archived HIV drug resistance mutations | 6 months
  Identify HIV drug resistance mutations in pro-viral HIV DNA

SECONDARY OUTCOMES:
HIV-1 reservoirs measurement | 1 year
  Quantification of pro-viral DNA

CONTACTS AND LOCATIONS:
Locations (1):
- Chantal Biya International Reference Centre, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: No
Participant data will be stored in a password protected computer